CLINICAL TRIAL: NCT03062761
Title: A Randomized, Controlled, Double Blind, Parallel Group, Multi-country Study to Investigate the Effects of an Infant Formula Containing Partially Hydrolysed Proteins on Growth, Safety and Tolerance in Healthy Term Infants
Brief Title: A Clinical Study to Investigate the Effects of an Infant Formula Containing Partially Hydrolysed Proteins on Growth, Safety and Tolerance in Healthy Term Infants
Acronym: TENUTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EBB15BL89832
Record Dates: First submitted 2017-02-03; First posted 2017-02-23 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Growth
MeSH Terms: interventions — Infant Formula; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active product: partially hydrolysed proteins (Experimental): Partially hydrolysed whey protein based infant formula containing prebiotics.
  Interventions: Other: Infant Formula with prebiotics
- Control product: standard formula (intact protein) (Active Comparator): Intact cow's milk protein based infant formula containing prebiotics.
  Interventions: Other: Standard Infant Formula

INTERVENTIONS:
Other: Infant Formula with prebiotics — Intervention group: Partially hydrolysed whey protein based infant formula containing prebiotics.
  Arms: Active product: partially hydrolysed proteins
Other: Standard Infant Formula — Control group: Intact cow's milk protein based infant formula containing prebiotics
  Arms: Control product: standard formula (intact protein)

SUMMARY:
It is universally accepted that the best nutrition for a new-born infant is breast milk. Breast milk provides a complete set of nutrients to support growth and development of children in early life, including components that have a beneficial effect on gut health and the body's ability to defend itself against infectious organisms and other invaders (immune system).However, it may occur that a mother is unable to breastfeed her child, or chooses not to breastfeed. In such cases, an infant formula inspired by breast milk is the best alternative. Research is done to optimize milk formula for infants. One of these formulas contains 'partially hydrolyzed' proteins instead of intact proteins, meaning the proteins in this formula are broken down into smaller pieces. These smaller pieces of protein make the milk more suitable for consumption by infants at risk of developing cow's milk allergy. These types of partially hydrolyzed protein formulas have been on the market for several years, in particular for children with a family risk of allergy. So far, no safety related issues have been reported. It is also known that weight gain of infants receiving partially hydrolyzed proteins in general is appropriate according to the World Health Organisation growth standards.

The main purpose of the TENUTO study is to demonstrate that infants who receive a specific partially hydrolyzed protein infant formula for the first 4 months of life have a similar weight gain compared to infants receiving standard infant formula with intact proteins. A group of infants who receive breast milk only is also included for comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy term infants (gestational age ≥ 37 weeks + 0 days and ≤ 41 weeks + 6 days);
2. Infants' age at enrolment ≤ 14 days;
3. Birth weight within normal range for gestational age and sex (10th to 90th percentile according to the WHO Child Growth Standards - or local growth standards if available);
4. Head circumference at inclusion within normal range for age and sex (within 2 SD curves according to WHO Child Growth Standards - or local growth standards if available);
5. Infant formula arms: infants who are exclusively formula fed by time of randomisation with a maximum infants' age of 14 days (infants of mothers who choose not to breastfeed or mothers who cease breastfeeding for any reason before the infant is 14 days of age); OR Breastfeeding reference arm: infants who are exclusively breastfed and whose mothers are intending to exclusively breastfeed their infant at least until the infant is 17 weeks of age; 6 Written informed consent from parent(s) and/or legal guardian(s) aged ≥ 18 years.

Exclusion Criteria:

Infants of pregnant women/mothers:

1. who are currently participating or will participate in any other (clinical) study involving investigational or marketed products during pregnancy and/or lactation;
2. known to have a significant medical condition (including during pregnancy) that might interfere with the study or known to affect intra-uterine growth (e.g. placenta previa, pre-eclampsia, eclampsia, gestational diabetes requiring insulin or oral medication), as per investigator's clinical judgement;

   Infants of parents:
3. who are incapable to comply with study protocol or Investigator's uncertainty about the willingness or ability of the parents to comply with the protocol requirements;

   Infants:
4. who have to be fed with a special diet other than standard (non-hydrolysed) cow's milk based infant formula
5. known to have current or previous illnesses/conditions which could interfere with the study or its outcome parameters, such as gastrointestinal malformations, congenital metabolic disorders, immune deficiency or major surgery, as per investigator's clinical judgement;
6. with any history of, or current participation in any other study involving investigational or marketed products.

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 380 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Weight gain | 17 weeks
  Weight gain in grams per day from baseline until 17 weeks of age

SECONDARY OUTCOMES:
Length | 17 weeks
  Gain in Recumbent length (mm/day)
Head circumference | 17 weeks
  Gain in Head circumference (mm/day)
Mid-upper arm circumference | 17 weeks
  Gain in Mid-upper arm circumference (mm/day)
Anthropometric measures | 17 weeks
  Z scores of anthropometric parameters
Albumin level | 17 weeks
  Albumin in blood (g/L)
Calcium level | 17 weeks
  Calcium in blood (mmol/l)
Phosphorus level | 17 weeks
  Phosphorus in blood (mmol/l)
Iron level | 17 weeks
  Iron (µmol/l) in blood
Magnesium level | 17 weeks
  Magnesium (mmol/l) in blood
Nitrogen level | 17 weeks
  Blood urea nitrogen (mmol/l)
Number of subjects with adverse events | 17 weeks
  Adverse events (by "System/Organ Class" and "Preferred term" according the MedDRA ) will be reported as number of subjects with at least one adverse event
Number of adverse events | 17 weeks
  Number of adverse events (by "System/Organ Class" and "Preferred term" according the MedDRA)
Concomitant medications | 17 weeks
  All concomitant medications (according to WHO-DDE) will be summarised in individual data listing
Regurgitation | 4, 8, 13 and 17 weeks
  Regurgitation nr of occurrences per week
Vomiting | 4, 8, 13 and 17 weeks
  Vomiting nr of occurrences per week
Diarrhoea | 4, 8, 13 and 17 weeks
  Number of infants with diarrhoea (definition adapted from WHO definition based on number of watery stools per day)
Constipation | 4, 8, 13 and 17 weeks
  Number of infants with constipation (definition adapted from Rome II criteria based on number of defecations and consistency per week)

CONTACTS AND LOCATIONS:
Locations (15):
- University of Turku Children's Allergy and Asthma Clinic, Turku, Finland
- France (2):
  - Groupement des Hopitaux de l'institut Catholique de Lille, Lille
  - Hospices Civils de Lyon, Lyon
- Germany (2):
  - Vivantes Klinik für Geburtsmedizin, Klinikum Neukölln, Berlin
  - Paediatric Practice, Bramsche
- Gelre Ziekenhuizen, Apeldoorn, Netherlands
- Poland (5):
  - Poliklinika Ginekologiczno-Poloznicza Sp. z o.o. Sp.k, Bialystok
  - Specjalistyczna Poradnia Medyczna Przylądek Zdrowia, Krakow
  - POLMED / Instytut Mikroekologii, Poznan
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - NZLA Michalkowice Jarosz i Partnerzy Spolka Lekarska, Siemianowice Śląskie
- Spain (4):
  - Hospital Quirónsalud Barcelona, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitari Sant Joan de Reus (IISPV), Reus
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: No